CLINICAL TRIAL: NCT03124459
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of ACE-083 in Patients With Charcot-Marie-Tooth Disease Types 1 and X
Brief Title: Study of ACE-083 in Patients With Charcot-Marie-Tooth Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: (Investigation of ACE-083 for use in patients with CMT is being discontinued as it did not achieve functional secondary endpoints in the A083-03 trial.
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A083-03; ACE-083 (Other: Acceleron Pharma Inc.)
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: CMT1 / CMTX
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth disease, X-linked, 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Cohort 1 (Experimental): ACE-083 150 mg intramuscular (IM) (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  Interventions: Drug: ACE-083
- Part 1 Cohort 2 (Experimental): ACE-083 200 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  Interventions: Drug: ACE-083
- Part 1 Cohort 3 (Experimental): ACE-083 up to 250 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  Interventions: Drug: ACE-083
- Part 2 (double-blind placebo controlled) (Experimental): ACE-083 up to 250 mg IM (tibialis anterior muscle) or placebo, once every 3 weeks for up to 9 doses
  Interventions: Drug: ACE-083; Drug: Placebo
- Part 2 (open label) (Experimental): ACE-083 up to 250 mg IM (tibialis anterior muscle), once every 3 weeks for up to 8 doses
  Interventions: Drug: ACE-083

INTERVENTIONS:
Drug: ACE-083 — Part 1 - Recombinant fusion protein. Part 2 - Recombinant fusion protein or buffer solution.
Drug: Placebo — Recombinant fusion protein or buffer solution
  Arms: Part 2 (double-blind placebo controlled)

SUMMARY:
This is a multicenter, phase 2 study to evaluate the safety, tolerability, pharmacodynamics (PD), efficacy, and pharmacokinetics (PK) of ACE-083 in patients with Charcot-Marie-Tooth Disease Type 1 and Type X (CMT1 and CMTX), to be conducted in two parts. Part 1 is non-randomized, open-label, dose-escalation and Part 2 is randomized, double-blind, and placebo-controlled.

DETAILED DESCRIPTION:
Part 1 (non-randomized, open-label, dose-escalation)

Part 1 will consist of up to 3 cohorts of 6 patients each and will evaluate multiple ascending dose levels of ACE-083 administered bilaterally once every 3 weeks for up to 5 doses in the tibialis anterior (TA) muscle. Patients in each cohort will be enrolled in a 4-week screening period before beginning treatment.

Part 2 (randomized, double-blind, placebo-controlled) Prior to the initiation of Part 2, a review of safety and efficacy data from Part 1 will be conducted by the Safety Review Team (SRT) to determine the recommended dose level (maximum 250 mg/muscle). A total of up to 40 new patients may be enrolled and randomized (1:1 randomization) to receive either ACE 083 (n=20) or placebo (n=20) bilaterally by injection into both TA muscles once every 3 weeks for up to 17 doses.

Study duration for Parts 1 and 2 for each patient will be approximately 24 weeks, including a 4-week screening period, a 12-week treatment period, and an 8-week follow-up period after the last dose.

Study duration for Part 2 will be 15 months, including 4-week screening, 6 months double blind placebo-controlled, 6 months open-label and 8 week follow-up.

ELIGIBILITY:
Key Inclusion Criteria

1. Age ≥ 18 years
2. Diagnosis of CMT1 or CMTX confirmed by:

   1. Clinical presentation and electrodiagnostics
   2. Genetically-confirmed CMT1 or CMTX for the patient or first-degree relative
3. Part 1:

   1. Six-minute walk distance (6MWD) of at least 150 meters (without a brace or walker)
   2. Independent ambulation for at least 10 meters, without a brace
   3. Left and right ankle plantar flexion MRC grade 4+ to 5, inclusive

   Part 2:
   1. 6MWD ≥ 150 and ≤ 500 meters (without a brace or walker); a maximum of 20% of enrolled patients with 6MWD ≥ 450 meters will be included
   2. Left and right ankle plantar flexion MRC grade 4- to 5, inclusive
4. Left and right ankle dorsiflexion Medical Research Council (MRC) manual muscle testing (MMT) grade 3 to 4+ inclusive. No more than 12 of the 40 subjects may have a grade of 3 or 3+ on one or both sides.
5. Females of childbearing potential must have negative urine pregnancy test prior to enrollment and use highly effective birth control methods during study participation and for 8 weeks following the last dose of ACE-083. Males must agree to use a condom during any sexual contact with females of childbearing potential while participating in the study and for 8 weeks following the last dose of ACE-083, even if he has undergone a successful vasectomy.
6. Ability to adhere to the study visit schedule/procedures, and to understand and comply with protocol requirements
7. Signed written informed consent

Key Exclusion Criteria

1. History of active malignancy, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
2. Symptomatic cardiopulmonary disease, significant functional impairment, significant orthopedic or neuropathic pain, or other co morbidities that in the opinion of the investigator would limit a patient's ability to complete strength and/or functional assessments on study
3. Type 1 or type 2 diabetes mellitus
4. Thyroid disorder unless condition is stable with no change in treatment for at least 4 weeks before the first dose and no expected change for duration of study
5. Renal impairment (serum creatinine ≥ 2 times the upper limit of normal (ULN])
6. Aspartate transaminase (AST) and/or alanine transaminase (ALT) ≥ 3 times ULN
7. Increased risk of bleeding (i.e., due to hemophilia, platelet disorders, or use of any anticoagulation/platelet modifying therapies up to 2 weeks prior to Study Day 1 and for duration of study; low dose aspirin [≤ 100 mg daily] is permitted)
8. Severe deformity or ankle fixation that would sufficiently limit passive range of motion to affect assessment of dorsiflexion strength
9. Major surgery within 4 weeks prior to Study Day 1
10. Chronic pharmacologic doses of systemic corticosteroids (≥ 2 weeks) within 4 weeks before Study Day 1 and for duration of study; intra-articular/topical/inhaled/intranasal physiologic doses of systemic corticosteroids are permitted
11. Androgens, growth hormone, insulin or oral hormone replacement therapy within 6 months before Study Day 1 and for duration of study; topical physiologic androgen replacement is permitted
12. Any change in medications potentially affecting muscle strength or function within 4 weeks of Study Day 1 and for duration of study (e.g., creatinine, CoQ10, systemic beta-adrenergic agonists)
13. Previous exposure to any investigational agent potentially affecting muscle volume, muscle strength, or muscle or nerve function within 5 half-lives of last dose plus an additional 8-week washout period (or 12 weeks prior to Study Day 1 if half-life is unknown)
14. Any previous or current exposure to ACE-083
15. Significant change in physical activity or exercise (e.g., significant increase or decrease in intensity or frequency) within 8 weeks before Study Day 1 or inability to maintain the baseline level of physical activity throughout the study
16. Any condition that would prevent MRI scanning or compromise the ability to obtain a clear and interpretable scan of the lower leg, as applicable (e.g., knee/hip replacement metallic implants)
17. Known active substance abuse, including alcohol
18. History of sensitivity to protein pharmaceuticals
19. Female that is lactating/breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Backstrom, MD, Study Chair — Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA
Locations (16):
- United States (16):
  - University of California-Irvine, Orange, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center - Neurology Department, Kansas City, Kansas
  - University of Minnesota, Neurology Department, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Neurology, Rochester, New York
  - Carolinas Healthcare System Neurosciences Institute, Charlotte, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomas FP, Brannagan TH 3rd, Butterfield RJ, Desai U, Habib AA, Herrmann DN, Eichinger KJ, Johnson NE, Karam C, Pestronk A, Quinn C, Shy ME, Statland JM, Subramony SH, Walk D, Stevens-Favorite K, Miller B, Leneus A, Fowler M, van de Rijn M, Attie KM. Randomized Phase 2 Study of ACE-083 in Patients With Charcot-Marie-Tooth Disease. Neurology. 2022 Jun 6;98(23):e2356-e2367. doi: 10.1212/WNL.0000000000200325. PMID 35545446

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Cohort 1 (150 mg): ACE-083 150 mg intramuscular (IM; tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 2 (200 mg): ACE-083 200 mg IM, (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 3 (240 mg): ACE-083 240 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 2 (Double-blind Placebo Controlled) Placebo Arm: Placebo once every 3 weeks for up to 9 doses
  ACE-083: Part 2 -buffer solution
- Part 2 (Double-blind Placebo Controlled) ACE-083 Arm: ACE-083 240 mg IM (tibialis anterior muscle) once every 3 weeks for up to 9 doses
  ACE-083: Part 2 - Recombinant fusion protein
- Part 2 (Open-label) ACE-083 Arm: ACE-083 240 mg IM (tibialis anterior muscle) once every 3 weeks for up to 8 doses
  ACE-083: Part 2 - Recombinant fusion protein
Period: Part 1-Open Label Dose Escalation
Arm/Group | Part 1 Cohort 1 (150 mg) | Part 1 Cohort 2 (200 mg) | Part 1 Cohort 3 (240 mg) | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm | Part 2 (Open-label) ACE-083 Arm
Started (Participants in the Part 2 double-blind placebo controlled portion of the study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 6 | 6 | 6 | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study. Participants that completed the double-blind portion of the study then moved into this Part 2 open-label portion of the study.)
Completed | 6 | 6 | 6 | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 0 (Patients in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study. Participants that completed the double-blind portion of the study then moved into this Part 2 open-label portion of the study.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2- Randomized Doubled-blind
Arm/Group | Part 1 Cohort 1 (150 mg) | Part 1 Cohort 2 (200 mg) | Part 1 Cohort 3 (240 mg) | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm | Part 2 (Open-label) ACE-083 Arm
Started (Participants in Part 1 Open-Label Dose escalation portion of the study were not the same participants that participated in the double-blind placebo controlled study.) | 0 (Participants in Part 1 Open-Label Dose escalation portion of the study were not the same participants that participated in the double-blind placebo controlled study.) | 0 (Participants in Part 1 Open-Label Dose escalation portion of the study were not the same participants that participated in the double-blind placebo controlled study.) | 0 (Participants in Part 1 Open-Label Dose escalation portion of the study were not the same participants that participated in the double-blind placebo controlled study.) | 21 (Participants in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 24 (Participants in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study.) | 0 (Participants in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study. Participants that completed the double-blind portion of the study then moved into this Part 2 open-label portion of the study.)
Completed | 0 | 0 | 0 | 9 | 5 | 0
Not Completed | 0 | 0 | 0 | 12 | 19 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 11 | 12 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 0
Period: Part 2- Open Label ACE-083
Arm/Group | Part 1 Cohort 1 (150 mg) | Part 1 Cohort 2 (200 mg) | Part 1 Cohort 3 (240 mg) | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm | Part 2 (Open-label) ACE-083 Arm
Started (Participants in Part 1 Open-Label Dose escalation portion of the study were not the same participants that participated in the double-blind placebo controlled study. Participants that completed the Part 2 double-blind placebo controlled portion of the study were able to move into the open-label portion of the study.) | 0 | 0 | 0 | 0 (Participants in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study. Participants that completed the double-blind placebo controlled portion of Part 2, moved into the open-label portion part 2 study.) | 0 (Participants in the double-blind placebo controlled study were not the same participants that participated in the Part 1 Open-Label Dose escalation portion of the study. Participants that completed the double-blind placebo controlled portion of Part 2, moved into the open-label portion part 2 study.) | 40 (The open-label portion of Part 2 are the participants that were enrolled in and completed the double-blind placebo-controlled portion of Part 2.)
Completed | 0 | 0 | 0 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 23
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all randomized patients who have received at least 1 dose of study drug (includes placebo). Additionally, the participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2. The open-label baseline measures are captured separately.
Groups:
- Part 1 Cohort 1: ACE-083 150 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 2: ACE-083 200 mg IM, (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 3: ACE-083 240 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 2 (Double-blind Placebo Controlled) Placebo: Placebo once every 3 weeks for up to 9 doses
  ACE-083: Part 2 - buffer solution.
- Part 2 (Double-blind Placebo Controlled) ACE-083: ACE-083 up to 250 mg IM (tibialis anterior muscle) once every 3 weeks for up to 9 doses
  ACE-083 Part 2 - Recombinant fusion protein
- Part 2 (Open-label) ACE 083-03 Arm: ACE-083 up to 250 mg IM (tibialis anterior muscle) once every 3 weeks for up to 8 doses
  ACE-083 Part 2 - Recombinant fusion protein
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 (Double-blind Placebo Controlled) Placebo | Part 2 (Double-blind Placebo Controlled) ACE-083 | Part 2 (Open-label) ACE 083-03 Arm | Total
Number analyzed (Participants) | 6 | 6 | 6 | 21 | 24 | 40 | 103
Age, Categorical [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2. The open-label baseline measures are captured separately.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 21 | 24 | 0 | 63
    <=18 years | 0 | 1 | 0 | 1 | 0 |  | 2
    Between 18 and 65 years | 6 | 5 | 6 | 17 | 23 |  | 57
    >=65 years | 0 | 0 | 0 | 3 | 1 |  | 4
Age, Categorical [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    <=18 years |  |  |  |  |  | 0 | 0
    Between 18 and 65 years |  |  |  |  |  | 36 | 36
    >=65 years |  |  |  |  |  | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient in the Phase 2 randomized portion of the study was randomized (to the ACE-083 arm) but not dosed.
  years
    number analyzed (Participants) | 6 | 6 | 6 | 21 | 23 | 0 | 62
    (all) | 40 (18.1) | 39 (17.8) | 49 (9.7) | 47.1 (15.3) | 45.8 (11.2) |  | 45.3 (13.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    (all) |  |  |  |  |  | 47.3 (12.9) | 47.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient in the Phase 2 randomized portion of the study was randomized (to the ACE-083 arm) but not dosed.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 21 | 23 | 0 | 62
    Female | 3 | 3 | 4 | 13 | 17 |  | 40
    Male | 3 | 3 | 2 | 8 | 6 |  | 22
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    Female |  |  |  |  |  | 28 | 28
    Male |  |  |  |  |  | 12 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient in the Phase 2 randomized portion of the study was randomized (to the ACE-083 arm) but not dosed.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 21 | 23 | 0 | 62
    Hispanic or Latino | 0 | 0 | 0 | 2 | 1 |  | 3
    Not Hispanic or Latino | 6 | 6 | 5 | 19 | 22 |  | 58
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    Hispanic or Latino |  |  |  |  |  | 3 | 3
    Not Hispanic or Latino |  |  |  |  |  | 37 | 37
    Unknown or Not Reported |  |  |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient in the Phase 2 randomized portion of the study was randomized (to the ACE-083 arm) but not dosed.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 21 | 23 | 0 | 62
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0
    Asian | 1 | 0 | 0 | 0 | 2 |  | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 |  | 0
    White | 5 | 6 | 6 | 21 | 20 |  | 58
    More than one race | 0 | 0 | 0 | 0 | 0 |  | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    American Indian or Alaska Native |  |  |  |  |  | 0 | 0
    Asian |  |  |  |  |  | 1 | 1
    Native Hawaiian or Other Pacific Islander |  |  |  |  |  | 0 | 0
    Black or African American |  |  |  |  |  | 0 | 0
    White |  |  |  |  |  | 38 | 38
    More than one race |  |  |  |  |  | 1 | 1
    Unknown or Not Reported |  |  |  |  |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2. The open-label baseline measures are captured separately.
  Participants
    United States: number analyzed (Participants) | 6 | 6 | 6 | 21 | 24 | 0 | 63
    United States | 6 | 6 | 6 | 21 | 24 |  | 63
Region of Enrollment [Number; unit: participants] — Population: The participants in the Open-Label portion of Part 2 are a sub-set of the participants that enrolled and then subsequently completed the double-blind placebo controlled portion of Part 2.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40
    United States |  |  |  |  |  | 40 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Frequency of Adverse Events
Description: Number of subjects with at least one adverse event related to treatment intervention from Part 1 of this study. Since this outcome measure was only pre-specified for Part 1, only data from the Part 1 participants is reported.
Time Frame: From initiation of treatment (Study Day 1) to end of follow-up period for Part 1 (Study Day 141).
Population: The Safety Set consists of all patients enrolled in the study who have received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Cohort 1 (150 mg): ACE-083 150 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
Arm/Group | Part 1 Cohort 1 (150 mg) | Part 1 Cohort 2 (200 mg) | Part 1 Cohort 3 (240 mg)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 6 | 5 | 6

2. Primary Outcome: Part 2: Percent Change in Muscle Volume to the End of the Double-blind Placebo-controlled Portion of the Study.
Description: The percent change from baseline in volume of injected muscle, by MRI compared to the Day 190 Assessment is reported. The pre-specified timepoint for this outcome was only for data collected from participants to the end of the double-blind placebo controlled portion of the study, therefore data for the open-label arm of the study is not reported.
Time Frame: From initiation of treatment (Study Day 1) to end of follow-up period of the double-blind placebo-controlled portion of the study (Study Day 190).
Population: Per Protocol Set: All participants enrolled/randomized in the study who received at least 1 dose of the study drug (includes placebo) with no major protocol violations
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 19
percent change | 2.2 (4.1) | 15.8 (4.3)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.01, ANCOVA; Mean Difference (Final Values) = 13.5, 90% CI 2-sided [4.9 to 22.1], Standard Error of Mean 5.2

3. Secondary Outcome: Part 2: Absolute Change in Amount of Intramuscular Fat Tissue to the End of the Double-blind Placebo-controlled Portion of the Study
Description: The absolute change from baseline in intramuscular fat fraction of the injected muscle, by MRI compared to Day 190 Assessment is reported. The pre-specified timepoint for this outcome was only for data collected from participants to the end of the double-blind placebo controlled portion of the study, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm3
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 19
mm3 | 1 (1.8) | -2.1 (1.9)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.16, ANCOVA; Mean Difference (Final Values) = -3.1, 90% CI 2-sided [-6.8 to 0.6], Standard Error of Mean 2.2

4. Secondary Outcome: Part 2: Percent Change in Muscle Strength to the End of the Double-blind Placebo-controlled Portion of the Study
Description: Percent change from baseline in strength of the injected muscle, by Quantitative Muscle Testing (QMT) compared to Day 190 Assessment is reported. The pre-specified timepoint for this outcome was only for data collected from participants to the end of the double-blind placebo controlled portion of the study, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 19 | 17
percent change | -3.4 (19.8) | 32.0 (19.8)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.13, ANCOVA; Mean Difference (Final Values) = 35.4, 90% CI 2-sided [-3.2 to 74], Standard Error of Mean 23.5

5. Secondary Outcome: Part 2: Percent Change in Muscle Function - Walk/Run Time to the End of the Double-blind Placebo-controlled Portion of the Study
Description: The percent change from baseline in functional assessments, as measured by 10-meter walk/run time when compared to Day 190 Assessment is reported. The pre-specified timepoint for this outcome was only for data collected from participants to the end of the double-blind placebo controlled portion of the study, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 19
Percent change | -10.1 (4.7) | -8.2 (4.7)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.73, ANCOVA; Mean Difference (Final Values) = 1.9, 90% CI 2-sided [-7.1 to 10.9], Standard Error of Mean 5.5

6. Secondary Outcome: Part 2: Percent Change in Muscle Function - Walk Distance Assessed at the End of the Double-blind Placebo-controlled Portion of the Study
Description: Percent change from baseline in functional assessments, as measured by 6-minute walk distance when compared to Day 190 Assessment, is reported. The pre-specified timepoint for this outcome was only for data collected from participants to the end of the double-blind placebo controlled portion of the study, therefore data for the open-label arm of the study is not reported.
Time Frame: From initiation of treatment (Study Day 1) to end of follow-up period for the double-blind placebo-controlled portion of the study (Study Day 190).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 19
Percent change | 6 (4) | 9.1 (3.8)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.51, ANCOVA; Mean Difference (Final Values) = 3.1, 90% CI 2-sided [-4.6 to 10.9], Standard Error of Mean 4.7

7. Secondary Outcome: Part 2: Change in Balance and Fall Risk at the End of the Double-blind Placebo-controlled Portion of the Study.
Description: Change from baseline in static and dynamic balance, as measured by the Berg Balance Scale, a 14-item scoring system to assess balance and fall risk in adults. The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. Total scores are used for reporting, with a range of 0-56, with higher scores mean a better demonstration of function. A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. The pre-specified timepoints for reporting are baseline Berg scale score and Day 190 score, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 20
score on scale
  Baseline | 52.8 (1.99) | 50.8 (5.58)
  Day 190 | 53 (2.77) | 51.4 (5.6)

8. Secondary Outcome: Part 2: Percent Change in Balance and Fall Risk From Baseline to the End of the Double-blind Placebo-controlled Portion of the Study
Description: Percent change was calculated for the difference from baseline and Day 190 Assessment scores on the Berg Balance Scale. The Berg Balance Scale, is a 14-item scoring system to assess balance and fall risk in adults. The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. Total scores are used for reporting, with a range of 0-56, with higher scores mean a better demonstration of function. A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. The pre-specified timepoints for reporting are baseline Berg scale score and Day 190 score, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in score on scale
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 20
percent change in score on scale | 0.4 (3.59) | 1.3 (3.13)

9. Secondary Outcome: Part 2: Change in Clinical Examination Score From Baseline to End of the Double-blind Placebo-controlled Portion of the Study
Description: Change from baseline in the Charcot-Marie-Tooth (CMT) Examination Score, version 2 (CMTES2), a composite scoring system to assess sensory and motor impairment in subjects with CMT. The total score is a subset of the following items from the CMT neuropathy score instrument: Sensory symptoms, Motor symptoms (legs), Motor symptoms (arms), Pinprick Sensibility, Vibration, Strength (legs), and Strength (arms). Each individual item is assessed using a rating from 0 to 4 inclusive. The range of CMTES2 scores is from 0 to 28 inclusive. A higher score means a greater degree of symptom severity. The Baseline score and score on the Day 190 Assessment are reported. The pre-specified timepoints for reporting are baseline Berg scale score and Day 190 score, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 20
score on scale
  Baseline | 10.1 (3.4) | 10.9 (3.67)
  Day 190 | 9.5 (3.02) | 11.2 (4.77)

10. Secondary Outcome: Part 2: Percent Change in Clinical Examination Score in Baseline to End of the Double-blind Placebo-controlled Portion of the Study
Description: Percent change was calculated for the difference in the Charcot-Marie-Tooth (CMT) Examination Score (CMTES2) from baseline and Day 190 Assessment scores. The pre-specified timepoints for reporting are baseline Berg scale score and Day 190 score, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in score on scale
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 20 | 20
percent change in score on scale | -0.2 (34.63) | 2.4 (24.26)

11. Secondary Outcome: Part 2: Change in Patient-reported Quality of Life From Baseline to the End of the Double-blind Placebo-controlled Portion of the Study
Description: The absolute change from baseline in Charcot-Marie-Tooth Health Index (CMT-HI), a disease-specific, patient-reported health index score from baseline and Day 190 Assessment scores. The pre-specified timepoints for reporting are baseline Berg scale score and Day 190 score, therefore data for the open-label arm of the study is not reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: absolute change in score on a scale
Arm/Group | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm
Number analyzed (Participants) | 19 | 18
absolute change in score on a scale | -0.2 (3.3) | -2.2 (3.1)
Statistical Analysis 1: Comparison: Part 2 (Double-blind Placebo Controlled) Placebo Arm vs Part 2 (Double-blind Placebo Controlled) ACE-083 Arm; Test type: Superiority; p = 0.63, ANCOVA; Mean Difference (Final Values) = -1.9, 90% CI 2-sided [-8.4 to 4.6], Standard Error of Mean 3.9

ADVERSE EVENTS:
Time Frame: Part 1 adverse events (AEs) were collected from baseline through Day 141. For Part 2, AEs were collected from on or after the first double-blind study drug administration up to the end of the double-blind period (Day 190). For the open-label period, adverse events are defined as AEs that started or worsened in intensity on or after the first open-label study drug administration up to the end of the study(Day 393/end-of-study).
Groups:
- Part 1 Cohort 1(150mg): ACE-083 150 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 2 (200mg): ACE-083 200 mg IM, (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 1 Cohort 3 (250mg): ACE-083 up to 250 mg IM (tibialis anterior muscle), once every 3 weeks for up to 5 doses.
  ACE-083: Part 1 - Recombinant fusion protein.
- Part 2 (Double-blind Placebo Controlled) Placebo Arm: Placebo, once every 3 weeks for up to 9 doses
  ACE-083:
  Part 2 - Placebo: buffer solution
- Part 2 (Double-blind Placebo Controlled) ACE-083 Arm: ACE-083 up to 250 mg IM (tibialis anterior muscle) once every 3 weeks for up to 9 doses
  ACE-083:
  Part 2 - Recombinant fusion protein
Arm/Group | Part 1 Cohort 1(150mg) | Part 1 Cohort 2 (200mg) | Part 1 Cohort 3 (250mg) | Part 2 (Double-blind Placebo Controlled) Placebo Arm | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm | Part 2 (Open Label)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/21 | 0/23 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 1/21 | 0/23 | 1/40
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 19/21 | 20/23 | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1(150mg) (N=6) | Part 1 Cohort 2 (200mg) (N=6) | Part 1 Cohort 3 (250mg) (N=6) | Part 2 (Double-blind Placebo Controlled) Placebo Arm (N=21) | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm (N=23) | Part 2 (Open Label) (N=40)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1(150mg) (N=6) | Part 1 Cohort 2 (200mg) (N=6) | Part 1 Cohort 3 (250mg) (N=6) | Part 2 (Double-blind Placebo Controlled) Placebo Arm (N=21) | Part 2 (Double-blind Placebo Controlled) ACE-083 Arm (N=23) | Part 2 (Open Label) (N=40)
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 4 | 6 | 8
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 2 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 7 | 6
joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 1
muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 6 | 6
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 1
limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
injection site discomfort (General disorders) | 3 | 2 | 3 | 4 | 4 | 4
injection site bruising (General disorders) | 2 | 2 | 2 | 1 | 6 | 6
injection site erythema (General disorders) | 2 | 1 | 1 | 1 | 7 | 10
injection site pain (General disorders) | 1 | 1 | 1 | 2 | 6 | 6
injection site swelling (General disorders) | 1 | 1 | 1 | 2 | 6 | 8
injection site pruritus (General disorders) | 1 | 0 | 1 | 0 | 5 | 6
injection site discoloration (General disorders) | 0 | 1 | 0 | 1 | 1 | 2
injection site macule (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
injection site warmth (General disorders) | 1 | 0 | 0 | 2 | 4 | 7
peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 2 | 3
fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
injection site dysaethesia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
injection site induration (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
injection site papule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
medical device site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2
nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2 | 3 | 4
upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1
viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
localised infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
pneunomia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3
conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 5 | 5 | 11
ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2
thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 5 | 3 | 7
skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1
arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 3
memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 2
restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0
burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1
dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 3
nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1
skin warm (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
gastrointestinal disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 3
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 3
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
rhinorrheoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 3
Behcet's syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
crystal urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
myoglobin blood increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
thyroxine free increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 4
bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
decreased appetitie (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 2
attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
inflammation of lacrimal passage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated because the statistically significant increase in total muscle volume (TMV) failed to translate to statistically significant improvements in functional or disease-related quality of life secondary endpoints in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03124459/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03124459/SAP_001.pdf